CLINICAL TRIAL: NCT02984904
Title: Multicenter Study About Fusarium Keratitits in Spain 2012 to 2014
Brief Title: Fusarium Keratitits in Spain 2012 to 2014
Status: Completed | Type: Observational
Sponsor: Miguel Armando Mosquera Gordillo, MD (Other)
Collaborators: Complejo Hospitalario de Navarra (Other)
Responsible Party: Sponsor-Investigator, Miguel Armando Mosquera Gordillo, MD, MD, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Other Study IDs: MMG-FUS-2015-01
Record Dates: First submitted 2016-11-17; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-11

CONDITIONS: Corneal Ulcer; Fusarium Infection
Keywords: Fusarium Infection; Corneal ulcer; Spain; Epidemiology
MeSH Terms: conditions — Corneal Ulcer; Fusariosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: survey — survey

SUMMARY:
The aim of this study was to describe the clinical-epidemiological characteristics of a series of cases of fungal keratitis associated with Fusarium spp., In Spain during the years 2012 to 2014.

DETAILED DESCRIPTION:
Corneal ulcers are the second cause of preventable blindness in tropical countries, which are produced by a wide variety of eye infections that can lead to visual impairment, As a consequence of the cicatrization of the lesions caused. The World Health Organization (WHO) estimates that around 1.5-2.0 million new cases of monocular blindness secondary to this type of lesions occur every year.

Corneal ulceration is attributed to mycotic aetiology between 6 and 53% of the cases, recognising at least 70 different genera. Studies in developing countries have reported the presence of a wide variety of pathogenic fungi isolated from corneal ulcers, most prominently highlighting Candida spp. And Aspergillus spp., however, the appearance of less common fungal pathogens, but of great medical importance, owing to increased morbidity in healthy patients and especially in the immunocompromised population. These pathogens include the filamentous fungi Fusarium spp.

Fusarium spp. Is a universally distributed opportunistic fungus, ubiquitous and of great economic importance because it is usually phytopathogenic. This fungus causes human infections such as keratitis, endophthalmitis, among others. A predisposing factor for Fusarium spp. Is the corneal trauma, with an incidence ranging from 7% to 89.9%. Some research shows that these lesions were caused by different agents, it includes plant material (rice, hawthorn, hay, among others), animal (insects, cat scratch, among others), dust, earth, mud, stones, glass, metal objects and nails. Other factors that affect the appearance of keratitis by this type of fungus include the use of topical corticosteroids, previous eye surgery, pre-existing eye diseases (lagophthalmos, chronic dacryocystitis, corneal scarring or corneal ulcer), systemic diseases such as diabetes mellitus, leprosy, among others. These mycotic infections tend to be resistant to conventional antifungal agents, presenting more severe complications than other types of infections.

The epidemiological pattern of Fusarium spp. keratitis varies from country to country, predominating in regions that share climatic conditions, as described in Florida, Ghana, and China. Even in one country, its distribution is not homogeneous, as evidenced by studies in southern India, between the years 1991 to 2000, where 1360 mycotic keratitis was present, 506 (37.2%) attributed to Fusarium spp. By contrast, a study conducted in northern India over 6 years found 61 cases of mycotic keratitis, 10 of them (16.4%) secondary to Fusarium spp.

In June 2006, the Centers for Disease Control and Prevention (CDC) confirmed an outbreak of Fusarium spp., In 164 patients with contact lenses in 33 states and 1 US territory, being the most important outbreak reported in this country.

The keratitis caused by Fusarium spp. Occurs infrequently in European countries with temperate climates. A study conducted in Paris between 1993 and 2001 reported 19 mycotic keratitis, 4 cases (21%) attributed to Fusarium spp.

In Spain, it has been realised clinical case studies of Fusarium spp, however, no descriptions of the epidemiological profile have been made.The aim of this study was to describe the clinical-epidemiological characteristics of a series of cases of fungal keratitis associated with Fusarium spp., In Spain during the years 2012 to 2014.

ELIGIBILITY:
Inclusion Criteria: Growth in the microbiological culture of Fusarium spp. In ocular samples informed by the participating centers confirmed or not by the National Center of Microbiology of the Carlos III Health Institute (ISC III) of Spain, admitting only one registry per patient / year -

Exclusion Criteria: Patients who could not be contacted because they did not reside in Spain or who did not accept the same

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Person diagnosed with keratitis secondary to Fusarium spp., During the study period
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Describe the clinical-epidemiological characteristics of a series of cases of fungal keratitis associated with Fusarium spp | 2012 to 2014
  epidemiological survey

CONTACTS AND LOCATIONS:
Overall Officials: José Larmarca Mateu, MD, Study Chair — CLINICA BARRAQUER; Tomas Marti Huguet, MD, Study Chair — HOSPITAL BELLVITGE; Sara Martin, MD, Study Chair — HOSPITAL UNIVERSITARIO VALL DE HEBRON; Paula Marticorena Alvarez, MD, Study Chair — Hospital Universitario La Princesa; Andres Garralda Luquin, MD, Study Chair — Complejo Hospitalario de Navarra; Carlos Lopez Gutierrez, MD, Study Chair — HOSPITAL GALDAKAO; Jesus Garrido Fierro, MD, Study Chair — HOSPITAL TXAGORRITXU - HOSPITAL UNIVERSITARIO ARABA; Raquel Feijó Lera, MD, Study Chair — HOSPITAL LAS CRUCES; Juan Carlos Sanchez España, MD, Study Chair — HOSPITAL GENERAL JUAN RAMÓN JIMENEZ; Graciela Trujillo, MD, Study Chair — HOSPITAL DOCTOR NEGRIN; Encarnacio Mengual Verdu, MD, Principal Investigator — Hospital Universitario San Juan de Alicante; Victor Garcia, MD, Study Chair — Hospital Universitario San Juan de Alicante; Miguel A Mosquera Gordillo, MD, Study Director — Hospital Universitario San Juan de Alicante; Natalia Baron Cano, Nurse, Study Chair — Miguel Hernandez University (MPH)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Upadhyay MP, Karmacharya PC, Koirala S, Tuladhar NR, Bryan LE, Smolin G, Whitcher JP. Epidemiologic characteristics, predisposing factors, and etiologic diagnosis of corneal ulceration in Nepal. Am J Ophthalmol. 1991 Jan 15;111(1):92-9. doi: 10.1016/s0002-9394(14)76903-x. PMID 1985498
- [Result] Ahearn DG, Zhang S, Stulting RD, Schwam BL, Simmons RB, Ward MA, Pierce GE, Crow SA Jr. Fusarium keratitis and contact lens wear: facts and speculations. Med Mycol. 2008 Aug;46(5):397-410. doi: 10.1080/13693780801961352. Epub 2008 Apr 4. PMID 18608899
- [Result] Whitcher JP, Srinivasan M, Upadhyay MP. Corneal blindness: a global perspective. Bull World Health Organ. 2001;79(3):214-21. Epub 2003 Jul 7. PMID 11285665
- [Result] Srinivasan M, Gonzales CA, George C, Cevallos V, Mascarenhas JM, Asokan B, Wilkins J, Smolin G, Whitcher JP. Epidemiology and aetiological diagnosis of corneal ulceration in Madurai, south India. Br J Ophthalmol. 1997 Nov;81(11):965-71. doi: 10.1136/bjo.81.11.965. PMID 9505820
- [Result] Bharathi MJ, Ramakrishnan R, Vasu S; Meenakshi; Palaniappan R. Aetiological diagnosis of microbial keratitis in South India - a study of 1618 cases. Indian J Med Microbiol. 2002 Jan-Mar;20(1):19-24. PMID 17657018
- [Result] Gopinathan U, Garg P, Fernandes M, Sharma S, Athmanathan S, Rao GN. The epidemiological features and laboratory results of fungal keratitis: a 10-year review at a referral eye care center in South India. Cornea. 2002 Aug;21(6):555-9. doi: 10.1097/00003226-200208000-00004. PMID 12131029
- [Result] Basak SK, Basak S, Mohanta A, Bhowmick A. Epidemiological and microbiological diagnosis of suppurative keratitis in Gangetic West Bengal, eastern India. Indian J Ophthalmol. 2005 Mar;53(1):17-22. doi: 10.4103/0301-4738.15280. PMID 15829742
- [Result] Norina TJ, Raihan S, Bakiah S, Ezanee M, Liza-Sharmini AT, Wan Hazzabah WH. Microbial keratitis: aetiological diagnosis and clinical features in patients admitted to Hospital Universiti Sains Malaysia. Singapore Med J. 2008 Jan;49(1):67-71. PMID 18204773
- [Result] Doczi I, Gyetvai T, Kredics L, Nagy E. Involvement of Fusarium spp. in fungal keratitis. Clin Microbiol Infect. 2004 Sep;10(9):773-6. doi: 10.1111/j.1469-0691.2004.00909.x. PMID 15355406
- [Result] Tanure MA, Cohen EJ, Sudesh S, Rapuano CJ, Laibson PR. Spectrum of fungal keratitis at Wills Eye Hospital, Philadelphia, Pennsylvania. Cornea. 2000 May;19(3):307-12. doi: 10.1097/00003226-200005000-00010. PMID 10832689
- [Result] Passos RM, Cariello AJ, Yu MC, Hofling-Lima AL. Microbial keratitis in the elderly: a 32-year review. Arq Bras Oftalmol. 2010 Jul-Aug;73(4):315-9. doi: 10.1590/s0004-27492010000400002. PMID 20944931
- [Result] Saha R, Das S. Mycological profile of infectious Keratitis from Delhi. Indian J Med Res. 2006 Feb;123(2):159-64. PMID 16575115
- [Result] Nath R, Baruah S, Saikia L, Devi B, Borthakur AK, Mahanta J. Mycotic corneal ulcers in upper Assam. Indian J Ophthalmol. 2011 Sep-Oct;59(5):367-71. doi: 10.4103/0301-4738.83613. PMID 21836342
- [Result] Green M, Apel A, Stapleton F. Risk factors and causative organisms in microbial keratitis. Cornea. 2008 Jan;27(1):22-7. doi: 10.1097/ICO.0b013e318156caf2. PMID 18245962
- [Result] Leck AK, Thomas PA, Hagan M, Kaliamurthy J, Ackuaku E, John M, Newman MJ, Codjoe FS, Opintan JA, Kalavathy CM, Essuman V, Jesudasan CA, Johnson GJ. Aetiology of suppurative corneal ulcers in Ghana and south India, and epidemiology of fungal keratitis. Br J Ophthalmol. 2002 Nov;86(11):1211-5. doi: 10.1136/bjo.86.11.1211. PMID 12386069
- [Result] Rosa RH Jr, Miller D, Alfonso EC. The changing spectrum of fungal keratitis in south Florida. Ophthalmology. 1994 Jun;101(6):1005-13. doi: 10.1016/s0161-6420(94)31225-5. PMID 8008340
- [Result] Xie L, Dong X, Shi W. Treatment of fungal keratitis by penetrating keratoplasty. Br J Ophthalmol. 2001 Sep;85(9):1070-4. doi: 10.1136/bjo.85.9.1070. PMID 11520759
- [Result] Chander J, Sharma A. Prevalence of fungal corneal ulcers in northern India. Infection. 1994 May-Jun;22(3):207-9. doi: 10.1007/BF01716706. PMID 7927819
- [Result] Chang DC, Grant GB, O'Donnell K, Wannemuehler KA, Noble-Wang J, Rao CY, Jacobson LM, Crowell CS, Sneed RS, Lewis FM, Schaffzin JK, Kainer MA, Genese CA, Alfonso EC, Jones DB, Srinivasan A, Fridkin SK, Park BJ; Fusarium Keratitis Investigation Team. Multistate outbreak of Fusarium keratitis associated with use of a contact lens solution. JAMA. 2006 Aug 23;296(8):953-63. doi: 10.1001/jama.296.8.953. PMID 16926355
- [Result] Rondeau N, Bourcier T, Chaumeil C, Borderie V, Touzeau O, Scat Y, Thomas F, Baudouin C, Nordmann JP, Laroche L. [Fungal keratitis at the Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts: retrospective study of 19 cases]. J Fr Ophtalmol. 2002 Nov;25(9):890-6. French. PMID 12515932
- [Result] Donnio A, Van Nuoi DN, Catanese M, Desbois N, Ayeboua L, Merle H. Outbreak of keratomycosis attributable to Fusarium solani in the French West Indies. Am J Ophthalmol. 2007 Feb;143(2):356-8. doi: 10.1016/j.ajo.2006.09.021. Epub 2006 Oct 20. PMID 17258535
- See also: Spectrum of Mycotic corneal ulcers in Mid Western peripheral region of Terrain belt of Nepal and Indo-Nepal Border — http://www.nepjol.info/index.php/NJMS/article/view/7651
- See also: Queratitis micótica. Caso clínico. Arch Soc Canar Oftal [Internet]. 2006;17 — http://www.oftalmo.com/sco/revista-21/21sco06.htm
- See also: Queratitis por Fusarium. A propósito de dos casos. Arch Soc Canar Oftal [Internet]. 2010;21 — http://www.oftalmo.com/sco/revista-21/21sco06.htm